CLINICAL TRIAL: NCT02886208
Title: Health Outcomes of Teens Participating in Summer Employment Immersion Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tamara S. Hannon, Associate Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1604487508
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Pediatric Obesity; Prediabetic State
MeSH Terms: conditions — Pediatric Obesity; Prediabetic State | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): This study has a single arm. All participants in a summer employment program at an urban farm in Indianapolis, IN are invited to participate.
  Interventions: Behavioral: Measurement

INTERVENTIONS:
Behavioral: Measurement — The intervention consists of diabetes prevention education sessions focusing on increasing physical activity and decreasing the intake of sugared drinks while increasing intake of fruits and vegetables. The 2-hr sessions occur weekly for 6 weeks. Height and weight is measured for each consenting participant at baseline and after 6 weeks. Participants are also asked to complete a short questionnaire to collect demographic and knowledge data. Outcome measures include: BMI, knowledge of physical activity and dietary habits conducive to diabetes prevention, and feelings of food insecurity.

SUMMARY:
This study is a collaboration between investigators and two community partners: a youth employment program and an urban farm. The community partners hire 300+ adolescents for summer jobs at various organizations. Approximately 120 adolescents will be employed with the urban farm site. As one component of their program evaluation plan, investigators will evaluate change in BMI of participants. The investigators hypothesize that there will be a reduction in BMI of those participants working at the urban farm site.

DETAILED DESCRIPTION:
The investigators will measure height/weight/BMI of all participants located at the urban farm site. Investigators will also collect demographic data as well as other social data (example: food security).

ELIGIBILITY:
Inclusion Criteria:

* employed by summer work program at urban farm

Exclusion Criteria:

* N/A

Ages: 15 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
BMI | 6 weeks

IPD SHARING:
Plan to Share IPD: No
Data will be published in a medical journal. There is no plan to make individual participant data available.